CLINICAL TRIAL: NCT00606021
Title: A Randomized Phase 2 Study Comparing Pemetrexed Plus Best Supportive Care With Best Supportive Care as Maintenance, Following First-Line Treatment With Pemetrexed-Cisplatin, in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study Comparing of Two Different Chemotherapy Regimens, in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11839; H3E-EZ-S114 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-17; First posted 2008-02-01 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

ARMS (2):
- A: Pemetrexed + Best Supportive Care (Experimental): Pemetrexed: 500 milligrams per square meter (mg/m²) , intravenous (IV), Day 1 of each 21-day cycle for 6 cycles
  Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
  Interventions: Drug: pemetrexed; Drug: Best Supportive Care
- B: Best Supportive Care (Active Comparator): Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
  Interventions: Drug: Best Supportive Care

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m², IV, Day 1 of each 21-day cycle for 6 cycles
  Other Names: Alimta; LY231514
  Arms: A: Pemetrexed + Best Supportive Care
Drug: Best Supportive Care — Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.

SUMMARY:
This is a multicenter, open-label, randomized, two-arm Phase 2 study comparing pemetrexed plus best supportive care with best supportive care alone as maintenance therapy following first-line treatment with a pemetrexed-cisplatin combination in patients with advanced non-squamous non-small cell lung cancer.

A total of approximately 100 patients are planned to be enrolled, and following completion of four cycles of pemetrexed-cisplatin (Induction Phase) those patients in which disease progression has not occurred will be randomized in a 2:1 ratio to one of two treatment arms (Maintenance Phase): Arm A (pemetrexed plus best supportive care) or Arm B (best supportive care alone).

ELIGIBILITY:
Inclusion criteria:

1. You must be at least 18 years old
2. You must have been diagnosed with non-squamous non-small cell lung cancer (NSCLC)
3. You must have had no prior systemic anticancer therapy for lung cancer
4. You must live close enough to the study doctor to be able to visit regularly for follow up
5. You must have signed informed consent form indicating your willingness to take part in this study
6. Your laboratory and medical history and tests must meet study requirements

Exclusion criteria:

1. Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
2. Prior radiotherapy and surgery should be completed at least 4 weeks prior to initiation of treatment
3. Serious concomitant systemic disorder (e.g., active infection including human immunodeficiency virus, or unstable cardiovascular disease)
4. Prior malignancy other than NSCLC, carcinoma in situ of the cervix, or nonmelanoma skin cancer unless treated at least 5 years previously with no subsequent evidence of recurrence
5. Brain metastasis
6. Presence of clinically significant (by physical exam) third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry
7. Significant weight loss (greater than 10%), over the previous 6 weeks before study entry
8. Concurrent administration of any other antitumor therapy
9. Inability to interrupt aspirin or other non-steroidal anti-inflammatory agents for a 5-day period (8-day period for long-acting agents such as piroxicam)
10. Inability or unwillingness to take folic acid, dexamethasone (or equivalent) or vitamin B12 supplementation
11. Pregnancy or breast-feeding
12. You are allergic to pemetrexed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9am to 5pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- Egypt (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asyut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mounofia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beirut, Lebanon
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Mubarak N, Gaafar R, Shehata S, Hashem T, Abigeres D, Azim HA, El-Husseiny G, Al-Husaini H, Liu Z. A randomized, phase 2 study comparing pemetrexed plus best supportive care versus best supportive care as maintenance therapy after first-line treatment with pemetrexed and cisplatin for advanced, non-squamous, non-small cell lung cancer. BMC Cancer. 2012 Sep 24;12:423. doi: 10.1186/1471-2407-12-423. PMID 23006447
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Induction phase (IP) is from first dose of study drug until randomization and entering to maintenance phase (MP) or discontinuation from treatment during IP. 106 participants were treated during IP. MP is from randomization to discontinuation from treatment. Overall period is IP+MP, whereas overall study is MP only.
Groups:
- Pemetrexed Plus Cisplatin (Induction Phase): Pemetrexed, 500 milligrams per square meter (mg/m²), intravenous (IV) followed by Cisplatin, IV, 75 mg/m² on Day 1 of each 21-day cycle for 4 cycles
- Pemetrexed Plus Best Supportive Care (Maintenance Phase): Pemetrexed: 500 (mg/m²), IV, Day 1 of each 21-day cycle for 6 cycles
  Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
- Best Supportive Care (Maintenance Phase): Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
Period: Induction Phase
Arm/Group | Pemetrexed Plus Cisplatin (Induction Phase) | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Started | 106 | 0 | 0
Completed | 19 | 0 | 0
Not Completed | 87 | 0 | 0
Not completed — Death | 73 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Period: Maintenance Phase
Arm/Group | Pemetrexed Plus Cisplatin (Induction Phase) | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Started | 0 | 28 | 27
Completed | 0 | 5 | 10
Not Completed | 0 | 23 | 17
Not completed — Death | 0 | 17 | 15
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pemetrexed Plus Best Supportive Care (Maintenance Phase): Pemetrexed: 500 mg/m², IV, Day 1 of each 21-day cycle for 6 cycles
  Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
- Total: Total of all reporting groups
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase) | Total
Number analyzed (Participants) | 28 | 27 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.52) | 62.9 (9.97) | 60.1 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 20 | 17 | 37
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 26 | 26 | 52
  African | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Egypt | 24 | 19 | 43
  Saudi Arabia | 0 | 1 | 1
  Lebanon | 4 | 7 | 11
Pathological Diagnosis [Number; unit: participants]
  Mixed Cell Carcinoma, Lung | 1 | 1 | 2
  Large Cells Lung Carcinoma | 8 | 5 | 13
  Adenocarcinoma | 19 | 21 | 40
Stage of Disease at The Time of Entry into This Study [Number; unit: participants]
  Stage III B - Locally advanced | 9 | 10 | 19
  Stage IV - Metastasized | 19 | 17 | 36
Eastern Cooperative Oncology Group (ECOG) Performance Status at randomization of maintenance phase [Number; unit: participants] — Classifies participants according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully active | 6 | 8 | 14
    1 - Ambulatory, restricted strenuous activity | 20 | 17 | 37
    2 - Ambulatory, unable to carry out work activity | 2 | 2 | 4
Lesion Response to induction phase [Number; unit: participants] — The lesions response is classified by the investigator according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. Complete Response (CR): disappearance of all target lesions; Partial Response: (PR) ≥30% decrease in sum of longest diameter of target lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD: ≥20% increase in sum of longest diameter of target lesions).
  participants
    Complete Response (CR) | 0 | 1 | 1
    Partial Response (PR) | 10 | 11 | 21
    Stable Disease (SD) | 17 | 13 | 30
    Unknown | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival During Maintenance Phase
Description: Progression free survival is defined as the time from randomization until the date of progression of disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD is ≥20% increase in sum of longest diameter of target lesions. PD in maintenance phase uses the last lesion assessment prior to randomization as the baseline assessment.
Time Frame: Randomization to progression of disease (PD) or date of death from any cause up to 30.9 months
Population: Participants who were randomized into maintenance phase and had measurable or evaluable lesions at baseline (last assessment before randomization) and post-baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Number analyzed (Participants) | 28 | 27
months | 3.2 [2.9 to 6.1] | 3.2 [2.2 to 4.3]
Statistical Analysis 1: Comparison: Pemetrexed Plus Best Supportive Care (Maintenance Phase) vs Best Supportive Care (Maintenance Phase); Test type: Superiority or Other; p = 0.1815, Regression, Cox — The significant level for the primary outcome measure of progression free survival during maintenance phase is one-sided 0.2; Stratified Cox regression model is used for hazard ratio estimate. Stratification factor: response status prior to randomization; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.42 to 1.37]

2. Secondary Outcome: Progression Free Survival During Overall Period (Induction Phase [IP] + Maintenance Phase [MP])
Description: Progression-free survival in overall period is defined as the time from the date of first dose of study drug during IP until the date of PD or death from any cause. PD was determined using RECIST criteria. PD is ≥20% increase in sum of longest diameter of target lesions. PD in overall period uses the screening lesion assessment prior to the induction phase as the baseline assessment.
Time Frame: First dose of study drug during IP to PD or date of death from any cause up to 33.6 months
Population: Participants who took at least one dose of study drug during IP and had measurable or evaluable lesions at baseline (assessment before induction phase) and post baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Number analyzed (Participants) | 28 | 27
months | 6.2 [6.0 to 8.3] | 6.0 [4.6 to 6.9]
Statistical Analysis 1: Comparison: Pemetrexed Plus Best Supportive Care (Maintenance Phase) vs Best Supportive Care (Maintenance Phase); Test type: Superiority or Other; p = 0.1233, Regression, Cox — The significant level for the secondary outcome measure of progression free survival during overall period is one-sided 0.2; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.40 to 1.26]

3. Secondary Outcome: Overall Survival During Maintenance Phase
Description: Overall survival in maintenance phase is defined as the time from randomization to death. Participants who were alive were censored at the last contact.
Time Frame: Randomization to PD or date of death from any cause up to 31.3 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Number analyzed (Participants) | 28 | 27
months | 12.2 [5.6 to 20.6] | 11.8 [6.3 to 25.6]
Statistical Analysis 1: Comparison: Pemetrexed Plus Best Supportive Care (Maintenance Phase) vs Best Supportive Care (Maintenance Phase); Test type: Superiority or Other; p = 0.7239, Regression, Cox — The significant level for the secondary outcome measure overall survival during maintenance period is two-sided 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.56 to 2.28]

4. Secondary Outcome: Overall Survival During Overall Period (IP + MP)
Description: Overall survival in overall period is defined as the time from first dose of study drug during IP to death. Participants who were alive were censored at the last contact.
Time Frame: First dose of study drug during IP to PD or date of death from any cause up to 34.1 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Number analyzed (Participants) | 28 | 27
months | 15.4 [8.4 to 23.7] | 16.4 [9.1 to 28.5]
Statistical Analysis 1: Comparison: Pemetrexed Plus Best Supportive Care (Maintenance Phase) vs Best Supportive Care (Maintenance Phase); Test type: Superiority or Other; p = 0.6376, Regression, Cox — The significant level for the secondary outcome measure overall survival during overall period is two-sided 0.05; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.59 to 2.38]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) During Overall Period
Description: The list of serious adverse events (SAEs) and other non-serious adverse events (AEs) are in Adverse Events Section.
Time Frame: First dose of study drug during IP through overall study completion (up to 34.3) months
Population: Participants who took at least one dose of study drug during IP, and randomized to maintenance phase.
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase) | Pemetrexed Plus Cisplatin (Induction Phase)
Number analyzed (Participants) | 28 | 27 | 106
participants
  Adverse Events (AE) | 15 | 16 | 74
  Serious Adverse Events (SAE) | 1 | 1 | 13

6. Secondary Outcome: Tumor Response Rate and Disease Control Rate After Induction Phase (IP)
Description: Tumor response rate (%) is the number of responders (participants with best response of CR or PR) divided by the number of participants qualified for tumor response according to RECIST criteria multiplied by 100. Disease control rate is percentage of participants with a best response of stable disease [SD], PR, or CR. CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; PD is≥20% increase in sum of longest diameter of target lesions. SD= neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Randomization to measured PD up to 31.4 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed Plus Best Supportive Care (Maintenance Phase) | Best Supportive Care (Maintenance Phase)
Number analyzed (Participants) | 28 | 27
percentage of participants
  Best Overall Response Rate | 0 [0.0 to 12.3] | 0 [0.0 to 12.8]
  CR | 0 [0 to 12.3] | 0 [0 to 12.8]
  PR | 0 [0.0 to 12.3] | 0 [0.0 to 12.8]
  SD | 57.1 [37.2 to 75.5] | 44.4 [25.5 to 64.7]
  Disease Control Rate | 57.1 [37.2 to 75.5] | 44.4 [25.5 to 64.7]
  PD | 32.1 [15.9 to 52.4] | 37.0 [19.4 to 57.6]
  Early Death From Malignant Disease | 7.1 [0.9 to 23.5] | 0 [0.0 to 12.8]
  Early Death From Toxicity | 0 [0.0 to 12.3] | 0 [0.0 to 12.8]
  Early Death From other cause | 3.6 [0.1 to 18.3] | 0 [0.0 to 12.8]
  Unknown | 0 [0.0 to 12.3] | 18.5 [6.3 to 38.1]

ADVERSE EVENTS:
Description: Adverse events include pre-existing conditions.
Groups:
- Pemetrexed Plus Best Supportive Care - Maintenance Phase: Pemetrexed: 500 mg/m², IV, Day 1 of each 21-day cycle for 6 cycles Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
- Best Supportive Care - Maintenance Phase: Best Supportive Care: Patients will receive best supportive care (dose, frequency, duration) as judged by their treating physician.
- Pemetrexed + Cisplatin - Induction Phase: Pemetrexed, 500 milligrams per square meter (mg/m²), intravenous (IV) followed by Cisplatin, IV, 75 mg/m² on Day 1 of each 21-day cycle for 4 cycles.
Arm/Group | Pemetrexed Plus Best Supportive Care - Maintenance Phase | Best Supportive Care - Maintenance Phase | Pemetrexed + Cisplatin - Induction Phase
Serious Adverse Events (participants affected / at risk) | 1/28 | 1/27 | 13/106
Other Adverse Events (participants affected / at risk) | 15/28 | 16/27 | 74/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Best Supportive Care - Maintenance Phase (N=28) | Best Supportive Care - Maintenance Phase (N=27) | Pemetrexed + Cisplatin - Induction Phase (N=106)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Best Supportive Care - Maintenance Phase (N=28) | Best Supportive Care - Maintenance Phase (N=27) | Pemetrexed + Cisplatin - Induction Phase (N=106)
Anaemia (Blood and lymphatic system disorders) | 5 (6) | 3 (3) | 14 (16)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (11) | 1 (1) | 11 (16)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 8 (10)
Nausea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 15 (20)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0) | 35 (65)
Chest pain (General disorders) | 4 (5) | 3 (3) | 8 (9)
Fatigue (General disorders) | 3 (3) | 4 (4) | 25 (30)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 26 (36)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 9 (9)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Due to a mistake in the randomization parameters form, the randomization was actually implemented in the ratio of 1:1 instead of the planned ratio of 2:1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days